CLINICAL TRIAL: NCT04407390
Title: Effects of Nicotinamide Riboside on the Clinical Outcome of Covid-19 in the Elderly. A Randomized Double-blind, Placebo-controlled Trial of Nicotinamide Riboside NR-COVID19
Brief Title: Effects of Nicotinamide Riboside on the Clinical Outcome of Covid-19 in the Elderly
Acronym: NR-COVID19
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No volunteers where recruited to this study. Other studies were prioritised over this at the time of enrollment.
Sponsor: University of Copenhagen (Other)
Collaborators: Bispebjerg Hospital (Other); Elysium Health (Industry)
Responsible Party: Principal Investigator, Morten Scheibye-Knudsen, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-20026601
Record Dates: First submitted 2020-05-22; First posted 2020-05-29 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: COVID
MeSH Terms: interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: Randomized double-blind case-control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Patients receiving placebo.
  Interventions: Dietary Supplement: Placebo
- NR (Experimental): Patients receiving nicotinamide riboside (NR-E)
  Interventions: Dietary Supplement: Nicotinamide riboside

INTERVENTIONS:
Dietary Supplement: Nicotinamide riboside — The patients will receive 1 g of nicotinamide riboside or placebo orally every morning for 14 days.
  Arms: NR
Dietary Supplement: Placebo — Placebo
  Arms: Control

SUMMARY:
The purpose of this study is to investigate whether nicotinamide riboside supplementation can attenuate the severity of SARS-CoV-2 infections in elderly patients.

A major event in aging is the loss of the central metabolite nicotinamide adenine dinucleotide (NAD+) that appear to be important in the proinflammatory environment that occur during aging. Notably, recent work from our and other groups suggest that aging can be ameliorated by even a short-term treatment of the NAD+ precursor nicotinamide riboside. Nicotinamide riboside has recently been shown to be able to return aging tissues to a younger state even after short term treatment. This vitamin B3- analog is naturally occurring, is readily taken up through oral administration and has been tested in human trials with few side effects. In this randomized double blinded case-control trial, the investigators will treat elderly (>70 year old) COVID19 patients with 1 g of nicotinamide riboside (NR-E) or placebo for 2 weeks and investigate if this affects the clinical course of the disease.

DETAILED DESCRIPTION:
Currently the number of SARS-CoV-2 positive patients are increasing worldwide and healthcare systems are attempting to cope with the massive pressure that this pandemic results in. Given the highly infectious virus and the relatively high mortality, this pandemic will likely result in many thousand casualties. Interventions are direly needed.

During the early reports of the pandemic it quickly became apparent that mortality was primarily attributed to the elderly population. Indeed, the mortality rate of young adults was around 0.2% while elderly Covid-19 patients displayed a mortality rate of ~20%. Thus, fatality rates increase ~100 fold when comparing young adults to elderly individuals.

A major event in aging is the loss of the central metabolite nicotinamide adenine dinucleotide (NAD+) that appear to be important in the proinflammatory environment that occur during aging. Notably, recent work from our and other groups suggest that aging can be ameliorated by even a short-term treatment of the NAD+ precursor nicotinamide riboside. Nicotinamide riboside has recently been shown to be able to return aging tissues to a younger state even after short term treatment. This vitamin B3- analog is naturally occurring, is readily taken up through oral administration and has been tested in human trials with few side effects. The purpose of this aim is to investigate if nicotinamide riboside can reduce the severity of COVID-19 in patients aged 70 or older.

The elderly population is particularly problematic because long term respirator use for these patients is connected with a substantial mortality risk. Interventions that can keep them from fulminant respiratory failure is therefore of critical importance.

1.2 Study treatment: Nicotinamide riboside Nicotinamide riboside (NR-E, supplied by Elysium Health) is a naturally occurring vitamin B3 analog produced by yeast and found in multiple food products at low concentration. Many organisms including humans cannot produce nicotinamide riboside but have evolved methods to convert this into the central redox modulator NAD+.

The efficacy and safety of nicotinamide riboside has been tested in a number of studies in both healthy controls and in patients suffering from metabolic disease, a risk factor for an adverse outcome of COVID-19 patients. Since this is a natural compound widely found in nature no subjects have yet developed allergic responses to the molecule, and repeated doses of up to 2 g orally per day have demonstrated an acceptable safety profile.

No treatment-emergent adverse events have so far been reported for nicotinamide riboside

1.3 Rationale NAD+ is emerging as a central metabolic molecule involved in multiple age-related pathways including inflammation and metabolic control. Notably, 2 weeks nicotinamide riboside treatment increases metabolic output, normalizes muscle function and reverses hypoxic responses in old mice. Recently, NAD+ has been shown to positively activate the inflammatory response in various tissue and may be involved in polarizing macrophages towards the M1 lineage and facilitate resolution of inflammation. Previously it was shown that SARS-CoV-1 evades activation of the immune response and exogenous activation of macrophages leads to a better outcome of SARS-CoV-1 infection. Thus, activation of elderly macrophages via NAD+ replenishment could be an efficacious strategy in COVID-19 patients. In addition, NAD+ replenishment may facilitate overall greater resilience of elderly patients considering the anti-aging effects of nicotinamide riboside allowing these patients to better cope with infections.

1.4 Rationale for study design and doses The purpose of this study is to investigate whether nicotinamide riboside supplementation can attenuate the severity of SARS-CoV-2 infections. The chosen dosage is 1 g per day given orally. This is lower than 2 g previously given to healthy elderly individuals, however, this particular patient population have not been treated with nicotinamide riboside previously so a slightly lower dose was chosen. In addition, there is data suggesting that NAD+ regulates circadian rhythm and the dose is therefore given in the morning.

The study design is as follows: Elderly patients (>70 years old) seen with suspected COVID-19 at Bispebjerg hospital that are not requiring oxygen therapy are subjected to a COVID-19 test. The patients will be asked if they want to participate in this trial. If the patients agree and if the COVID-19 test is positive the patients will be randomized to either placebo or 1g nicotinamide riboside daily. Previous work has shown an efficacious increase in NAD+ levels combined with better physiological outcomes after 2 weeks treatment in preclinical trials. The investigators will therefore treat patients for 2 weeks total with a primary outcome of the study being hypoxic respiratory failure as defined by needing oxygen therapy. The patients will be evaluated in the ambulatory at day 7 and after the treatment ends at day 14. Follow up in the ambulatory will occur three months after enrollment. If a patient is admitted to the hospital during the treatment period the treatment continues for the full two weeks. To evaluate outcomes, untargeted metabolomics and the NAD-ome will be measured in peripheral blood mononucleated cells (PBMCs) upon enrolment, at day 7 and immediately after the study as well as at follow up three months later. Changes in the epigenetic landscape is a strong biomarker of age and is affected by NAD+ and epigenetic evaluation will be performed in the PBMCs. Next generation machine learning data analysis will be applied to identify predictors of clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age 70 or older, inclusive at the time of diagnosis.
3. Body mass index between 18-40 kg/m2 (both inclusive) and weight ≥ 40 kg at enrolment.
4. A diagnosis of Covid-19.

Exclusion Criteria:

1. Need for oxygen therapy.
2. Ongoing severe acute respiratory syndrome.
3. Cancer diagnosis within last 5 years.
4. Unwillingness or inability to follow the procedures outlined in the protocol.
5. Concurrent enrollment in another clinical study involving an investigational treatment.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Hypoxic respiratory failure | Day 1
  Hypoxic respiratory failure as defined by need for oxygen therapy
Hypoxic respiratory failure | Day 7
  Hypoxic respiratory failure as defined by need for oxygen therapy
Hypoxic respiratory failure | Day 14
  Hypoxic respiratory failure as defined by need for oxygen therapy
Hypoxic respiratory failure | Day 90
  Hypoxic respiratory failure as defined by need for oxygen therapy

SECONDARY OUTCOMES:
Mortality | Day 1
  Overall mortality
Mortality | Day 7
  Overall mortality
Mortality | Day 14
  Overall mortality
Mortality | Day 90
  Overall mortality
Sepsis | Day 1
  Sepsis
Sepsis | Day 7
  Sepsis
Sepsis | Day 14
  Sepsis
Sepsis | Day 90
  Sepsis
Circulatory failure | Day 1
  Circulatory failure as defined by a need for interventions to support the circulatory system.
Circulatory failure | Day 7
  Circulatory failure as defined by a need for interventions to support the circulatory system.
Circulatory failure | Day 14
  Circulatory failure as defined by a need for interventions to support the circulatory system.
Circulatory failure | Day 90
  Circulatory failure as defined by a need for interventions to support the circulatory system.
Days in hospital | Day 1
  Days in hospital
Days in hospital | Day 7
  Days in hospital
Days in hospital | Day 14
  Days in hospital
Days in hospital | Day 90
  Days in hospital
NAD levels | Day 1
  Measurements of NAD+ and related metabolite levels by mass spectrometry in whole blood.
NAD levels | Day 7
  Measurements of NAD+ and related metabolite levels by mass spectrometry in whole blood.
NAD levels | Day 14
  Measurements of NAD+ and related metabolite levels by mass spectrometry in whole blood.
NAD levels | Day 90
  Measurements of NAD+ and related metabolite levels by mass spectrometry in whole blood.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: Undecided